CLINICAL TRIAL: NCT00382369
Title: Whole Genome Scan of Extended Families With Familial Vocal Cord Paralysis
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Kerem Eithan, Professor, Hadassah Medical Organization
Other Study IDs: VOCALCORD-HMO-CTIL
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Vocal Cord Paralysis
Keywords: familial vocal cord paralysis; genetic screening
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA prepared from blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Vocal cord paralysis is a common cause of congenital stridor and airway obstruction. In this study we plan to identify the genetic locus of the genes in two extended families who suffer of the disease.

DETAILED DESCRIPTION:
In a number of families suffering of familial vocal cord paralysis it has previously been shown that the disease is inherited autosomal dominant. In one of the families the gene coding for the disease was located on chromosome 6q16. We will be analyzing 2 extended families with familial vocal cord paralysis to define their genetic defect leading to the disease. All family members will undergo a laryngoscopy to determine the extent of paralysis. For all family members we will isolate DNA and determine their microsatellite polymorphism on chromosome 6q16. If the results are negative we will continue the study and perform a whole genome scan to localize the gene(s) involved.

ELIGIBILITY:
Inclusion Criteria:

* members of families suffering of familial vocal cord paralysis

Exclusion Criteria:

* none

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families suffering of familial vocal cord paralysis
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2008-11-17 (Actual); Study Completion 2008-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Kerem, MD, Study Director — Hadassah MO; Batsheva Kerem, PhD, Principal Investigator — Hebrew University Jerusalem
Locations (1):
- Hadassah-Hebrew University Medical Center, Mt Scopus, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manaligod JM, Skaggs J, Smith RJ. Localization of the gene for familial laryngeal abductor paralysis to chromosome 6q16. Arch Otolaryngol Head Neck Surg. 2001 Aug;127(8):913-7. doi: 10.1001/archotol.127.8.913. PMID 11493198